CLINICAL TRIAL: NCT06723366
Title: Protective Effect of Angong Niuhuang Against Negative Inflammatory Response and Neurologic Dysfunction After Cardiovascular Surgery (PANDA X)
Brief Title: Protective Effect of Angong Niuhuang Against Negative Inflammatory Response and Neurologic Dysfunction After Cardiovascular Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator of Department of Cardiovascular Surgery, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PANDA X
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Cardio-pulmonary Bypass; Cardiovascular Surgery; Cerebral Protection; Brain Injury
Keywords: Inflammatory Response; cardiopulmonary bypass
MeSH Terms: conditions — Brain Injuries | interventions — Angong Niuhuang Pill

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ANP group (Experimental)
  Interventions: Drug: Angong Niuhuang Pill (ANP)
- Control (Other): standard treatment
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Drug: Angong Niuhuang Pill (ANP) — Angong Niuhuang Pill (ANP) (3 g/pill, 1 pill/day for 5 days)
  Arms: ANP group
Other: Control (Standard treatment) — Blank control
  Arms: Control

SUMMARY:
Neurologic Dysfunction is one of the main factors contributing to poor outcomes in cardiac surgery patients, except for heart failure. Atherosclerosis of the aorta, a history of cerebral infarction, and cervical artery disease are common clinical risk factors for cerebral neurological dysfunction after cardiac surgery. Results of preclinical studies suggested that Angong Niuhuang Pills (ANPs), a traditional Chinese patent medicine, including realgar, cinnabaris, Bovis Calculus, artificial Moschus, and powdered buffalo horn extract, decreased infarct volume and cerebral edema, and presented anti- atherosclerosis and cardio-protective effects in clinical and preclinical studies. The PANDA X trial is designed as a pilot study to explore the safety and efficacy of ANP in patients with moderate-to-severe neurologic dysfunction after cardiovascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* (1) an age > 18 years,
* (2) underwent cardiovascular surgery,
* (3) diagnosis of acute neurologic dysfunction, including but not limited acute cerebral infarction of the internal carotid artery system,
* (4) a National Institutes of Health Stroke Scale (NIHSS) score ranging from 10 to 20,
* (5) a time from symptom onset to randomization within 36 h,
* (6) provision of informed consent.

Exclusion Criteria:

* (1) not suitable for taking ANP after the dialectical process by a traditional Chinese medical doctor,
* (2) received ANP within 1 month before stroke onset,
* (3) liver failure,
* (4) declined to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
changes in the NIHSS score | after 14 days of randomization
  a National Institutes of Health Stroke Scale (NIHSS) score ranging from 10 to 20

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li S, Wang A, Shi L, Liu Q, Guo X, Liu K, Wang X, Li J, Zhu J, Wu Q, Yang Q, Zhuang X, You H, Feng F, Luo Y, Li H, Ni J, Peng B. Safety and efficacy of Angong Niuhuang Pills in patients with moderate-to-severe acute ischemic stroke (ANGONG TRIAL): A randomized double-blind placebo-controlled pilot clinical trial. Chin Med J (Engl). 2025 Mar 5;138(5):579-588. doi: 10.1097/CM9.0000000000003133. Epub 2024 Nov 6. PMID 39501831